CLINICAL TRIAL: NCT02337595
Title: Transfusion of CD45RA-depleted Donor Lymphocytes to Improve Regeneration of Antimicrobial Immunity After TCR-alpha/Beta Depleted Hematopoietic Stem Cell Transplantation
Brief Title: Memory T-cell Infusion to Improve Immunity After TCR-alpha/Beta Depleted Hematopoietic Stem Cell Transplantation
Acronym: 45RA_NEG_DLI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CD45RA_NEG_DLI_2014FRCPHOI
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Immune Deficiency Disease; Bone Marrow Failure Syndromes; Opportunistic Infections; Graft vs Host Disease
Keywords: CD45RA-depletion; TCR-alpha/beta depletion; Hematopoietic Stem Cell Transplantation; immune reconstitution; Graft Enhancement, Immunologic; Immunocompromized Host
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Immune Deficiency Disease; Bone Marrow Failure Disorders; Opportunistic Infections; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: CD45RA-depleted peripheral blood mononuclear cells — Infusion of escalating doses of CD45RA-depleted donor-derived allogeneic peripheral blood mononuclear cells

SUMMARY:
The stud will evaluate whether infusions of CD45RA-depleted lymphocytes from the donor early post-transplant is a safe way to improve immunity to common infections in recipients of TCR-alpha/beta depleted hematopoietic stem cell grafts.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) remains the most important direct complication of hematopoietic stem cell transplantation. Methods used to prevent GVHD include diverse pharmacologic interventions and ex vivo methods of T-cell depletion, the latter being the most effective ones. Historically depletion of T-cells from the graft is associated with increased rate of graft failure, relapse of malignant disease and prolonged immune deficiency. Selective depletion of TCR-alpha/beta T-lymphocytes is a new method of hematopoietic stem cell graft manipulation which is thought to conserve important cell populations, e.g. NK cells and gamma/delta T cells within the graft. Preliminary results suggest that TCR alpha/beta depletion ensures high engraftment rate, low early mortality and good control of GVHD. The problem of delayed immune reconstitution and life-threatening viral infections remains incompletely resolved.

Depletion of naive (CD45RA-positive) T-cells was developed as a new method of graft manipulation to prevent GVHD. Research data indicate that alloreactivity is associated mainly with naive T-cell fraction. In vitro depletion of CD45RA lowers significantly the alloreactive response while retaining reactivity to pathogens.

In the current protocol we plan to test whether relatively low doses of CD45RA-depleted mononuclear cells can be safely infused after TCR-alpha/beta depleted transplantation. The biologic readout for the protocol will be quantitative assessment of T-cell reactivity to common pathogens after infusion.

ELIGIBILITY:
Inclusion Criteria:

* recipient of allogeneic hematopoietic stem cell graft from haploidentical or matched unrelated donor
* TCR alpha/beta depletion of the hematopoietic stem cell graft
* CMV-seropositive donor
* stable hematopoietic engraftment

Exclusion Criteria:

* active graft-versus-host disease grade 2-4
* any systemic immune suppressive therapy except calcineurin inhibitor monotherapy
* uncontrolled sepsis

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of grade 2-4 acute graft-versus-host disease | 100 days
  Cumulative incidence (competing risk model) of acute graft-versus-host disease
Immune reconstitution (Quantitative evaluation of lymphocyte subsets in the peripheral blood, quantitative evaluation of pathogen-specific immune response by ELISPOT assay) | 120 days
  Quantitative evaluation of lymphocyte subsets in the peripheral blood, quantitative evaluation of pathogen-specific immune response by ELISPOT assay

SECONDARY OUTCOMES:
1-year survival | 1 year
  Kaplan-Meyer estimate of overall survival
Transplant-related mortality | 1-year
  Cumulative incidence (competing risk model) of transplant-related mortality
Incidence of chronic graft-versus-host disease | 1 year
  Cumulative incidence (competing risk model) of chronic graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maschan, MD, Principal Investigator — Fedaral Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Federal Research Center for pediatric hematology, oncology and immunology, Moscow, Russia

REFERENCES:
- [Background] Teschner D, Distler E, Wehler D, Frey M, Marandiuc D, Langeveld K, Theobald M, Thomas S, Herr W. Depletion of naive T cells using clinical grade magnetic CD45RA beads: a new approach for GVHD prophylaxis. Bone Marrow Transplant. 2014 Jan;49(1):138-44. doi: 10.1038/bmt.2013.114. Epub 2013 Aug 12. PMID 23933765
- [Background] Bleakley M, Heimfeld S, Jones LA, Turtle C, Krause D, Riddell SR, Shlomchik W. Engineering human peripheral blood stem cell grafts that are depleted of naive T cells and retain functional pathogen-specific memory T cells. Biol Blood Marrow Transplant. 2014 May;20(5):705-16. doi: 10.1016/j.bbmt.2014.01.032. Epub 2014 Feb 11. PMID 24525279